CLINICAL TRIAL: NCT03184688
Title: The Long-term Effect of Platelet-rich Plasma in Patients With Carpal Tunnel Syndrome: a Prospective Randomized Double-blind Controlled Trial
Brief Title: Platelet Rich Plasma for Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yung-Tsan Wu, Attending Physician of Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Perineural PRP for CTS
Record Dates: First submitted 2017-06-07; First posted 2017-06-14 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Carpal Tunnel Syndrome
Keywords: platelet rich plasma; Perineural injection therapy; hydrodissection
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- platelet rich plasma injection (Experimental): The platelet rich plasma (PRP) is a new and potential treatment for peripheral neuropathy in many animal studies.
  Interventions: Procedure: platelet rich plasma
- Normal saline (Placebo Comparator): Normal saline for hydrodissection
  Interventions: Drug: Normal saline

INTERVENTIONS:
Procedure: platelet rich plasma — Ultrasound-guided PRP injection between proximal carpal tunnel and median nerve.
  Arms: platelet rich plasma injection
Drug: Normal saline — Ultrasound-guided normal saline injection between proximal carpal tunnel and median nerve.
  Arms: Normal saline

SUMMARY:
Carpal tunnel syndrome (CTS) is the most common peripheral entrapment neuropathy with involving compression of the median nerve in the carpal tunnel. Although many conservative managements of CTS, the effectiveness of these methods is insignificant or only persist for a short duration. The platelet rich plasma (PRP) is a new and potential treatment for patients with kinds of musculoskeletal disorders and recent reports showed being beneficial for peripheral neuropathy in animal studies. Since 2014, four small clinical trials showed the positive effect of PRP in peripheral neuropathy. Among these studies, two small trials showed beneficial effect of PRP for patients with mild CTS. However, the definite clinical effect of PRP for peripheral neuropathy from currently published studies is unclarified because these studies enrolled a few patients and lacked long-term follow-up (no more than 6 months follow-up).

DETAILED DESCRIPTION:
After obtaining written informed consent, patients of clinically diagnosed with bilateral CTS were randomized into intervention and control side. Intervention group received one-dose ultrasound-guided PRP injection and control group received one-dose ultrasound-guided normal saline injection. No additional treatment after injection through the study period. The primary outcome is Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) and secondary outcomes include visual analog scale (VAS), cross-sectional area (CSA) of the median nerve, sensory nerve conduction velocity of the median nerve, and finger pinch strength. The evaluation was performed pretreatment as well as on the 2nd week, 1st, 3rd, 6th month and one year after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-80 year-old.
* Diagnosis was confirmed using an electrophysiological study

Exclusion Criteria:

* Cancer
* Coagulopathy
* Pregnancy
* Inflammation status
* Polyneuropathy, brachial plexopathy
* Thoracic outlet syndrome
* Previously undergone wrist surgery or steroid injection for CTS

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline of pain on 2nd week, 1st, 3rd, 6th month and one year after the treatment. | Baseline, 2nd week, 1st, 3rd, 6th month and one year after treatment.
  Boston carpal tunnel syndrome questionnaire (BCTQ) is a frequently used patient-based questionnaire for measurement of carpal tunnel syndrome which encompasses symptom severity and functional status. Each question ranges from 1 to 5 with a higher score indicating severer symptom or a higher degree of disability. Total score ranges from 19 to 95 and the mean of total scores divided with each item score were used for further analysis.

SECONDARY OUTCOMES:
Change from baseline in severity of symptoms and functional status on 2nd week, 1st, 3rd, 6th month and one year after the treatment. | Baseline, 2nd week, 1st, 3rd, 6th month and one year after treatment.
  Using the Visual analog scale (VAS) to measure the pain scale before treatment and multiple time frame after treatment.
Change from baseline in cross-sectional area of the median nerve on 2nd week, 1st, 3rd, 6th month and one year after the treatment. | Baseline, 2nd week, 1st, 3rd, 6th month and one year after treatment.
  Using the musculoskeletal sonogram to measure the cross-sectional area of the median nerve.
Change from baseline in conduction velocity, amplitude of median nerve on 2nd week, 1st, 3rd, 6th month and one year after the treatment. | Baseline, 2nd week, 1st, 3rd, 6th month and one year after treatment.
  The antidromic sensory nerve conduction velocity of the median nerve was performed on all subjects according to the protocol reported by the American Academy of Neurology (USA). The median nerve was stimulated at the wrist between the palmar longus and flexor carpal radialis tendon at a distance of approximately 14 cm from the active electrode.
Change from baseline in finger pinch on 2nd week, 1st, 3rd, 6th month and one year after the treatment. | Baseline, 2nd week, 1st, 3rd, 6th month and one year after treatment.
  The finger pinch strength was measured using dynamometer (Fabrication Enterprises Inc., USA). The subject was seated with shoulder adducted and neutrally rotated with the elbow flexed at 90°. The forearm and wrist were positioned in a neutral position for the palmar pinch

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Tsan Wu, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Locations (1):
- Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital, Taipei, Neihu District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wu YT, Ho TY, Chou YC, Ke MJ, Li TY, Huang GS, Chen LC. Six-month efficacy of platelet-rich plasma for carpal tunnel syndrome: A prospective randomized, single-blind controlled trial. Sci Rep. 2017 Dec;7(1):94. doi: 10.1038/s41598-017-00224-6. Epub 2017 Mar 7. PMID 28273894
- [Result] Malahias MA, Johnson EO, Babis GC, Nikolaou VS. Single injection of platelet-rich plasma as a novel treatment of carpal tunnel syndrome. Neural Regen Res. 2015 Nov;10(11):1856-9. doi: 10.4103/1673-5374.165322. PMID 26807124
- [Result] Uzun H, Bitik O, Uzun O, Ersoy US, Aktas E. Platelet-rich plasma versus corticosteroid injections for carpal tunnel syndrome. J Plast Surg Hand Surg. 2017 Oct;51(5):301-305. doi: 10.1080/2000656X.2016.1260025. Epub 2016 Dec 6. PMID 27921443
- [Result] Mulvaney SW. Ultrasound-guided percutaneous neuroplasty of the lateral femoral cutaneous nerve for the treatment of meralgia paresthetica: a case report and description of a new ultrasound-guided technique. Curr Sports Med Rep. 2011 Mar-Apr;10(2):99-104. doi: 10.1249/JSR.0b013e3182110096. PMID 21623291